CLINICAL TRIAL: NCT03339882
Title: The Effect of Remifemin in Preventing the Climacteric Symptoms Caused by LHRH-a Treatment in Breast Cancer: a Randomized II-stage Clinic Research
Brief Title: Remifemin Preventing the Climacteric Symptoms in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-RICH1; 2017ZA030 (Other Grant/Funding Number: Zhejiang Program of Traditional Chinese Medicine)
Record Dates: First submitted 2017-10-15; First posted 2017-11-13 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Effect of Drugs; Safety Issues
Keywords: remifemin; preventive effect; LHRH-a; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Remifemin; black cohosh root extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifemin intervention (Experimental): Using Remifemin during LHRH-a treatment in breast cancer
  Interventions: Drug: Remifemin
- Control (No Intervention): No intervention during LHRH-a treatment in breast cancer

INTERVENTIONS:
Drug: Remifemin — Remifemin 0.2g po bid*12 weeks at the beginning of the LHRH-a treatment
  Other Names: cimicifuga racemosa; black cohosh
  Arms: Remifemin intervention

SUMMARY:
LHRH-a is an important hormone treatment in breast cancer especially in high-risk hormone receptor-positive patients or hormone receptor-negative but needing ovarian function protecting. The climacteric symptoms caused by LHRH-a are often and prominent, which is a common clinical problem.

DETAILED DESCRIPTION:
Ovarian function suppression (OFS) or protection has been studied widely in breast cancer. As an common drug in clinic, LHRH-a is an important method for OFS in breast cancer especially in high-risk hormone receptor-positive patients or hormone receptor-negative but needing ovarian function protecting. The climacteric symptoms caused by LHRH-a are often and prominent, which is a common clinical problem. Remifemin (cimicifuga racemosa / black cohosh) is effective in climacteric symptoms as a hormone replacement treatment, some research concluded that it is also safe in breast cancer patients who are postmenopausal or taking tamoxifen suffering from climacteric symptoms. While in China, more than 2/3 breast cancer patients are pre/peri-menopause, and some part of them should take OFS as an hormone treatment. OFS can cause sever climacteric symptoms in a short time. The investigators aim to estimate the effect and safety of Remifemin in climacteric symptoms caused by OFS in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. provision of informed consent
2. clinical stage I~IIIC
3. histologically proven invasive breast cancer
4. women defined as premenopausal according to NCCN guideline
5. plan to accept the LHRH-a as endocrine treatment or ovarian function protection

Exclusion Criteria:

1. clinical evidence of metastatic disease
2. bilateral oophorectomy
3. patients who, for whatever reason (e.g., confusion, infirmity, alcoholism), are unlikely to comply with trial requirements
4. patients who accepted anti-cancer treatment before
5. previous hormonal therapy as adjuvant treatment for non-cancer disease
6. patients unwilling to stop taking any drug known to affect sex hormonal status, or in whom it would be inappropriate to stop previous history of invasive malignancy within the last 5 years, other than squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix, adequately cone biopsied
7. treatment with a non-approved or experimental drug during 1 month before entry into the study
8. history of bleeding diathesis (i.e., Disseminated intravascular coagulation, clotting factor deficiency), or long term anticoagulant therapy (other than antiplatelet therapy and low dose warfarin)
9. leukopenia and/or thrombocytopenia
10. history of ocular fundus diseases
11. history of thromboembolic diseases
12. history of osteoporotic fractures

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Kupperman Item (KMI) | 3 months after treatment
  Scoring according to Kupperman item scale (Total: 0-48, the score higher the symptoms are severer) which includes of hot flash, sweat, insomnia, anxious, depressed, vertigo, fatigue, arthralgia, headache, palpitate (each item has a weighting coefficient according to four grade scores: no symptom *0, sometimes *1, always *2, influent life *3).

SECONDARY OUTCOMES:
Disease free survival | 2 years
  Disease free survival rate in 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xingfei Yu, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang C, Huang Q, Liang CL, Zhang YW, Deng DH, Yu Y, Chen DB, Yang HJ, Yu XF. Effect of cimicifuga racemosa on menopausal syndrome caused by LHRH-a in breast cancer. J Ethnopharmacol. 2019 Jun 28;238:111840. doi: 10.1016/j.jep.2019.111840. Epub 2019 Mar 29. PMID 30935866